CLINICAL TRIAL: NCT06996444
Title: Évaluation d'un Programme de santé du Pied Incorporant Des Chaussures Minimalistes Sur Les Facteurs de Risque de Chute Chez Des Personnes âgées Vivant en EHPAD : Une étude Pilote
Brief Title: Evaluation of a Foot Health Program Incorporating Minimalist Footwear on Fall Risk Factors in Older People Living in Senior Nursing Homes: a Pilot Study.
Acronym: GRAND'PAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RIPH2-FUNDENBERGER-GRAND'PAS; 2025-A00124-45 (Other: ANSM)
Record Dates: First submitted 2025-05-05; First posted 2025-05-30 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Fall Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Workshops to improve the mobility of the older people through foot health (Experimental): Study participants will benefit from a plantar massage session (5-10 min foot massage) and one posture and walking workshop per week, supervised by a trained health professional. Minimalist shoes have been purchased by the centers and used during the workshops.
  Interventions: Other: Program Including Various Workshops aiming to preserve elderly's autonomy through foot health

INTERVENTIONS:
Other: Program Including Various Workshops aiming to preserve elderly's autonomy through foot health — Combination of minimalist footwear, foot massages, and workshops to re-learn walking and posture

SUMMARY:
Every year in France, 2 million falls by people over 65 are responsible for 10,000 deaths, the leading cause of accidental death, and more than 130,000 hospitalizations.

The main objective of this study is to evaluate the evolution of mobility in older people living in nursing homes, following 12 foot health workshops, carried out by a health professional, including the wearing of minimalist shoes.

DETAILED DESCRIPTION:
The program is divided into 3 parts :

1. Foot preparation phase (1st to 3rd week): Study participants will receive one individual session per week of plantar massage (approximately 10 min massage), combined with foot stimulation exercises.
2. Transition phase (weeks 4 to 6): Study participants will benefit from a workshop of around 1 hr per week focusing on foot mobility, posture and walking. Minimalist shoes will be introduced and certain exercises will be performed with them. The shoes will be given to participants free of charge.
3. Stabilization phase (weeks 7 to 12): Study participants will benefit from the same foot health workshops with minimalist shoes. The shoes will also be left with the participants outside the workshops, so that they can use them independently.

ELIGIBILITY:
Inclusion Criteria:

* People over 65 years of age
* Able to walk independently with or without a walking aid (cane, walker, etc.)
* Persons affiliated with a social security system or assimilated
* Persons (participants, guardians, or curators where applicable) who have been informed and have given their written consent to participate in the study.

Exclusion Criteria:

* People who already wear minimalist shoes.
* People with a contraindication to wearing minimalist shoes
* People wearing orthopedic shoes prescribed by a health professional.
* People taking part in a falls prevention program.
* Persons unable to walk
* Persons with any other contraindication at the investigator's discretion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
the evolution of mobility | Before and immediatly after the program
  Timed up and go test

SECONDARY OUTCOMES:
The distance of the center of gravity from the center | Before the intervention (baseline) , immediatly after the intervention, and 12 weeks following the end of the intervention
  The stabilometry platform
Strength of the toes | Before the intervention (baseline) , immediatly after the intervention, and 12 weeks following the end of the intervention
  By dynamometer
Ankle joint amplitudes in dorsal flexion and plantar extension | Before the intervention (baseline) , immediatly after the intervention, and 12 weeks following the end of the intervention
  With a goniometer
Fear of falling | Before the intervention (baseline) , immediatly after the intervention, and 12 weeks following the end of the intervention
  Numerical scale from 0 to 10
Pain felt in the feet during ambulation | Before the intervention (baseline) , immediatly after the intervention, and 12 weeks following the end of the intervention
  Numerical scale from 0 to 10
Participants' satisfaction with the minimalist shoes | Before the intervention (baseline) , immediatly after the intervention, and 12 weeks following the end of the intervention
  Questionnaire
Number of hours shoes used | Immediately after intervention and 12 weeks after the end of the intervention
  Questionnaire
Fall | Immediately after intervention and 12 weeks after the end of the intervention
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Ehpad les Cèdres, Beaux
  - Ehpad Paradis, Espaly-Saint-Marcel
  - Ehpad Le Vergé de Léa, Le Puy-en-Velay
  - Ehpad Nazareth, Le Puy-en-Velay
  - Ehpad Saint Joseph, Le Puy-en-Velay

IPD SHARING:
Plan to Share IPD: Yes
Primary and secondary outcomes, demographic data
Supporting Information: Study Protocol